CLINICAL TRIAL: NCT02546687
Title: Prediction of Anastomotic Leak/Stricture After Esophagectomy With Gastric Pull-up by Venous Blood Gas
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Veacheslav Zilbermints, MD, Rabin Medical Center
Other Study IDs: 0251-15-RMC
Record Dates: First submitted 2015-08-09; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Esophagectomy
Keywords: Anastomotic Leak; Esophagectomy Gastric Pull-up
MeSH Terms: conditions — Anastomotic Leak | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood gas mesurment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Canidate for elective esophagectomy: Venous blood sampling from gastric tube during elective esophagectomy
  Interventions: Other: Venous blood sampling

INTERVENTIONS:
Other: Venous blood sampling — The investigators will take 1-2 cc of venous blood from proximal part of stomach before gastric tube creation and in the same time the investigators will take same amount of venous blood from peripheral vein. This blood will be analyzed in the "ABL800 FLEX blood gas analyzer" as a routine blood analyses that making by anesthesiologist during the operation. This blood sampling the investigators will make again after 15-30 minutes from the same area in proximal stomach (after creation of gastric tube) and peripheral vein just before anastomosis creation. The investigators will measure components of venous blood gases (O2, pH, CO2, lactate) from the area of future anastomosis before construction of gastric tube and just before creation of anastomosis ( after 15-30 minutes), compare the results of this analysis with systemic venous blood.

SUMMARY:
Esophageal resection becomes a routine surgical procedure in many medical centers. Usually reconstruction after esophagectomy is achieved by gastric pull-up with cervical or intrathoracic anastomosis. The only blood supply for this gastric tube is by right gastroepiploic arcade. Bad or borderline perfusion of gastric tube is the main reason for future anastomotic leaks or strictures.

The investigators suggest to measure components of venous blood gases (O2, pH, CO2, lactate) from the area of future anastomosis before construction of gastric tube and just before creation of anastomosis ( after 15-30 minutes), compare the results of this analysis with systemic venous blood.

The investigators suppose that elevation of acid features of blood (pH decreasing, lactate increasing etc.) as expression of tissue ischemia after gastric tube creation maybe the significant predictive sign for future anastomotic leaks or strictures.

After operation the investigators plan to find relationship between the blood gas changes and rate of anastomotic leak and stricture.

This is prospective study. Anticipated cohort of 50 patients

DETAILED DESCRIPTION:
Prediction of Anastomotic Leak/Stricture after Esophagectomy with Gastric Pull-up by Venous Blood Gas.

Esophageal resection becomes a routine surgical procedure in many medical centers. Usually reconstruction after esophagectomy is achieved by gastric pull-up with cervical or intrathoracic anastomosis. The only blood supply for this gastric tube is by right gastroepiploic arcade. Bad or borderline perfusion of gastric tube is the main reason for future anastomotic leaks or strictures.

There are a lot of methods for intraoperative assessment of gastric tube perfusion. This methods include basic (as color, temperature of tube) and advanced assessment as optical fiber spectroscopy, visible light spectroscopy, the combination of a laser Doppler flowmeter and spectrophotometer, a laser Doppler imager, partial tissue oxygen pressure with a Clark-type polar graphic oxygen electrode, continuous measurement of mucosal PCO2 using recirculation gas analysis with a TONOCAP device together with mean arterial pressure measurement, and cardiac output and systemic vascular resistance by pulse contour analysis laser-assisted fluorescent-dye angiography (1-5).

All this methods are comparative complicated and do not promise good assessment results.

The investigators suggest to measure components of venous blood gases (O2, pH, CO2, lactate) from the area of future anastomosis before construction of gastric tube and just before creation of anastomosis ( after 15-30 minutes), compare the results of this analysis with systemic venous blood.

The investigators suppose that elevation of acid features of blood (pH decreasing, lactate increasing etc.) as expression of tissue ischemia after gastric tube creation maybe the significant predictive sign for future anastomotic leaks or strictures.

After operation the investigators plan to find relationship between the blood gas changes and rate of anastomotic leak and stricture.

Objectives The aims of this study is to compare the changes in venous blood gas in gastric tube together with systemic venous blood before construction of gastric tube and just before creation of anastomosis . After operation the investigators plan to find relationship between the blood gas changes and rate of anastomotic leak and stricture.

Study Design This is prospective study. Anticipated cohort of 50 patients The investigators are planning to take 1-2 cc of venous blood from proximal part of stomach before gastric tube creation and in the same time the investigators will take same amount of venous blood from peripheral vein. This blood will be analyzed in the "ABL800 FLEX blood gas analyzer" (Radiometer Copenhagen) as a routine blood analyses that making by anesthesiologist during the operation. This blood sampling the investigators will make again after 15-30 minutes from the same area in proximal stomach (after creation of gastric tube) and peripheral vein just before anastomosis creation. Important that because of technical needs (regardless our study) this stomach area from where the investigators are going to get blood for analyses will be removed immediately after anastomosis creation. So there is no danger for future injury or tissue changes for the patient due to needle stubbing for blood analyses.

Every patient will undergo routine follow up in the surgical department for minimum 7-10 hospitalization days with describing signs of anastomotic leak. Patients will continue routine follow up in our outpatient clinic (as every patient after such kind of surgery) two weeks, 6 weeks and 3 months after discharge from surgical department with evaluation of anastomotic stricture signs.

Participants. Inclusion criteria Patients who scheduled to undergo elective esophagectomy with gastric pull-up reconstruction in Beilinson hospital and are willing and able to give inform consent.

Data collection and statistical analysis. Data will be collected about patients demographic data, comorbidities, kind of pathology, neoadjuvant treatment (for cancer patients), time of surgery, patient hemodynamic state during surgery. The investigators will collect blood results especially measure of O2, pH, CO2, lactate. After surgery the investigators will describe and collect clinical and radiological signs of anastomotic leak and stricture.

Statistical analysis. Logistic regression and ROC (receiver operating characteristic) will be used to assess relationship between the blood gas changes and rate of anastomotic leak and stricture.

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled to undergo elective esophagectomy with gastric pull-up reconstruction in Beilinson hospital and are willing and able to give inform consent.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who scheduled to undergo elective esophagectomy with gastric pull-up reconstruction in Beilinson hospital and are willing and able to give inform consent.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Criteria for defining a surgical site infection (SSI) | 3 months
  Data from: Mangram AJ, Horan TC, Pearson ML, et al. Guideline for prevention of surgical site infection. In: Infection Control and Hospital Epidemiology, CDC 1999; 20:247.
The Clavien-Dindo Classification of Surgical Complications | 3 months
  Ann of Surg 2009;250: 187-196
Definition and measurement of anastomotic leak | 3 months
  Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Bruce J1, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Br J Surg. 2001 Sep;88(9):1157-68.
Assessment of anastomotic stricture severity | 3 months
  Assessment of anastomotic stricture severity for minimal, mild, moderate, or severe by dysphagia assessment with standardized dysphagia severity score (Endoscopic and symptomatic assessment of anastomotic strictures following esophagectomy and cervical esophagogastrostomy. Williams VA1, Watson TJ, Zhovtis S, Gellersen O, Raymond D, Jones C, Peters JH. Surg Endosc. 2008 Jun;22(6):1470-6. Epub 2007 Nov 20.)
Assessment of anastomotic stricture severity | 3 months
  Assessment of anastomotic stricture severity by size for minimal (12 mm), mild (9-12 mm), moderate (5-8 mm), or severe (<5 mm) using endoscopy or Barium esophagram.